CLINICAL TRIAL: NCT06555341
Title: The Effect of Training Given With Three Different Models on the Skill of Nursing Students in Administering Insulin: Mix Methods
Brief Title: Insulin Administration Skills of Nursing Students
Acronym: Skills
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, AYSE SOYLU, Principal Investigator, Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: KahramamarasSIU
Record Dates: First submitted 2024-08-05; First posted 2024-08-15 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Diabetes Mellitus
Keywords: Six Thinking Hats; Video; Diabetes mellitus; Insulin; Training; Nursing
MeSH Terms: conditions — Diabetes Mellitus; Insulin Resistance

STUDY DESIGN:
Intervention Model Description: This research was designed as a mixed methods study. This type of methodology with the use of strong aspects of both quantitative and qualitative methods was selected to be able to discover different perspectives and determine relationships between complex layers of the research questions (Shorten & Smith, 2017). The study was conducted as a randomised, controlled study at the quantitative stage and a descriptive phenomenonological design was used at the qualitative stage. The reporting of the study followed the guidelines of the "Control List for the Development of Mixed Methods Research Methodology" (Fetters & Molina-Azorin, 2019).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Six Thinking Hats Group (Experimental): Six Thinking Hats Group
  Interventions: Behavioral: Experimental: Six Thinking Hats Group
- Video Group (Other): Video Group
  Interventions: Behavioral: Other: Video Group
- Control Group (No Intervention): Control Group

INTERVENTIONS:
Behavioral: Experimental: Six Thinking Hats Group — 2. Subcutaneous insulin administration was explained with the traditional training model.
  3. The Six Thinking Hats technique and how it is used was then explained in detail to the students. Any points that were not fully understood were explained again so that the technique was thoroughly reinforced.
  4. The researchers had made hats from different coloured card. All the students wore all the hats in turn and were asked the questions related to that colour hat as stated above (semi-structured questionnaire 1-6).
  5. The responses given by the students to the questions were audio-recorded. Each interview lasted 30 mins.
  Arms: Six Thinking Hats Group
Behavioral: Other: Video Group — 2. Subcutaneous insulin administration was explained with the traditional training model.
  3. Then by scanning the QR code from the nursing practice skills textbook(Aylaz & Yakıncı, 2024), the researchers provided the link for the students to watch the insulin application video.
  4. Without mentioning hat colours or the Six Thinking Hats method to this group, the questions on the semi-structured questionnaire were asked, and the interviews, each lasting 30 mins, were audio-recorded.
  5. After completing the video training, the mid-test data were collected by applying the Subcutaneous Insulin Application Skill Level Observation Form during administration of insulin to a dummy.
  Arms: Video Group

SUMMARY:
Aim: The effects of training delivered to nursing students through the traditional method, the Six Thinking Hats method, and the video method were examined on insulin application skill.

Method: This study, using mixed methods was conducted between 15 February and 15 May 2024, with a total sample of 90 nursing students. The control group (n=30) received traditional training only. The Six Thinking Hats group (n=30) received traditional training and Six Thinking Hats training. The video group (n=30) received traditional training and video training. Three skill measurements were taken at the same times from all the groups. The video and Six Thinkng Hats groups were asked open-ended questions and the responses were recorded. Quantitative data were analyzed using IBM SPSS vn.23 software and qualitative data with MAXQDA 2024.

DETAILED DESCRIPTION:
To increase the knowledge and procedural skills of nursing students and avoid incorrect applications, the aim of this multi-dimensional study was to measure the effect on the insulin application skill of students given training in insulin administration with the traditional learning model, the video model, and the Six Thinking Hats model. In accordance with these aims, the following hypotheses were tested; H11: The Six Thinking Hats learning model would have an effect on the skill of nursing students in administering subcutaneous insulin.

H12:. The video learning model would have an effect on the skill of nursing students in administering subcutaneous insulin.

METHOD Study Design This research was designed as a mixed methods study. This type of methodology with the use of strong aspects of both quantitative and qualitative methods was selected to be able to discover different perspectives and determine relationships between complex layers of the research questions . The study was conducted as a randomised, controlled study at the quantitative stage and a descriptive phenomenonological design was used at the qualitative stage. The reporting of the study followed the guidelines of the "Control List for the Development of Mixed Methods Research Methodology" .

Study Sample Power analyis was performed based on a sample in literature, and it was calculated that there should be 20 participants in each of the three groups to provide an effect size of d=1.2119816, α err prob=0.05, and power (1-β err prob)=0.95 . In consideration of potential losses during the study, it was planned to include 30 subjects in each group, and thus the study was completed with a total of 90 nursing students (Figure 1, CONSORT diagram). To ensure data saturation, the purposeful sampling method was used at the qualitative stage .

Study Inclusion Criteria • Nursing students who were willing to participate in the study, completed all the stages of the study process, and had not received any previous insulin application training.

Study Exclusion Criteria

• Not meeting the study inclusion criteria in full. Randomisation and Blinding A computer program producing random numbers was used in the randomisation process (http://www.randomizer.org/form.htm). Using the randomisation list, the students were randomly assigned to the video group, the Six Thinking Hats group, or the control group according to the class list. As the students did not know the groups, a single blinded technique was used .

Study Variables Independent Variables The Six Thinking Hats model or the video watched by the experimental groups together with some sociodemographic characteristics.

Dependent Variables The mean subcutaneous insulin application skill points of the students. Data Collecion Tools The study data were collected using a Personal Information Form, a Subcutaneous Insulin Application Skill Level Observation Form, and a Semi-Structured questionnaire.

Personal Information Form:

This sociodemographic information form was formed of 3 questions related to age, gender, and status of having previously received insulin application training .

Subcutaneous Insulin Application Skill Level Observation Form:

This form, measures the skill of subcutaneous insulin administration. The form consists of 13 items and the content validity index has been calculated as 0.92 (>0.64) . The Cronbach alpha coefficient obtained in this study was 0.90.

Semi-structured Questionnaire:

For each of the six different coloured hats, the nursing students were asked questions as follows:

1. For the white hat referring to neutrality and objectivity; what knowledge do you have about insulin pen application? How did you obtain this information?
2. For the red hat referring to emotions and subjectivity; How is the insulin treatment process of the patient affected when hand hygiene is not followed when administering insulin and the date of the insulin is not checked?
3. For the yellow hat referring to clarity and positivity; what is the benefit to the patient of clockwise rotation when administering insulin? Why is it important to leave a space of 1cm between one application and the next? Why do we expel ½ unit of insulin before administration?
4. For the black hat referring to caution and risk assessment; if insulin is not adminisered according to the 10 correct principles, what type of complications can develop? What may happen if you discard the needle tip covered with the small cap and not the large cap after the application?
5. For the green hat referring to creative ideas; what innovative teaching models do you think could be used for insulin application training to be more consolidated and permanent?
6. For the blue hat referring to process control; what have you learned so far about insulin application? What have you gained from the insulin application training?

Data Collection Six Thinking Hats Group

1. The pre-test data of the experimental group students were collected by applying the Subcutaneous Insulin Application Skill Level Observation Form during administration of insulin to a dummy.
2. Subcutaneous insulin administration was explained with the traditional training model.
3. The Six Thinking Hats technique and how it is used was then explained in detail to the students. Any points that were not fully understood were explained again so that the technique was thoroughly reinforced.
4. The researchers had made hats from different coloured card. All the students wore all the hats in turn and were asked the questions related to that colour hat as stated above (semi-structured questionnaire 1-6).
5. The responses given by the students to the questions were audio-recorded. Each interview lasted 30 mins.
6. After finishing recording the responses to the Six Thinking Hats questions, the Subcutaneous Insulin Application Skill Level Observation Form was applied during administration of insulin to a dummy, and the mid-test data were collected.
7. At 3 months after the Six Thinking Hats training, the final test data were collected by applying the Subcutaneous Insulin Application Skill Level Observation Form during administration of insulin to a dummy.

Video Group

1. The pre-test data of the video group students were collected by applying the Subcutaneous Insulin Application Skill Level Observation Form during administration of insulin to a dummy.
2. Subcutaneous insulin administration was explained with the traditional training model.
3. Then by scanning the QR code from the nursing practice skills textbook , the researchers provided the link for the students to watch the insulin application video.
4. Without mentioning hat colours or the Six Thinking Hats method to this group, the questions on the semi-structured questionnaire were asked, and the interviews, each lasting 30 mins, were audio-recorded.
5. After completing the video training, the mid-test data were collected by applying the Subcutaneous Insulin Application Skill Level Observation Form during administration of insulin to a dummy.
6. At 3 months after the video training, the final test data were collected by applying the Subcutaneous Insulin Application Skill Level Observation Form during administration of insulin to a dummy.

Control Group

1. The pre-test data of the control group students were collected by applying the Subcutaneous Insulin Application Skill Level Observation Form during administration of insulin to a dummy.
2. Subcutaneous insulin administration was explained with the traditional training model.
3. After completing the traditional training, the mid-test data were collected by applying the Subcutaneous Insulin Application Skill Level Observation Form during administration of insulin to a dummy.
4. At 3 months after the traditional training, the final test data were collected by applying the Subcutaneous Insulin Application Skill Level Observation Form during administration of insulin to a dummy.

Statistical Analysis Content analysis was used in the interpretation of qualitative data. The students were asked semi-structured questions in face-to-face interviews and the responses were audio recorded. These recorded interviews were decoded by the researchers through repeated listenings. After the decoding, data analysis was performed with a process of code-category-theme analysis. Methodologically, the inductive coding path was followed in the data analysis . Max Qualitative Data Analysis (MAXQDA) Analytics Pro2024 program was used in the analysis. Qualitative analysis was performed by the first author and the other two authors examined the analyses to ensure the highest data quality. The analyses were thus overseen and confirmed according to the accuracy of the notes of each of the authors. This stage confirmed the data coding and ensured reliability. In this way the reliability of the study was tested through the suitability, transferability, reliability, credibility, and rigour of the data collected .

The quantitative data of the study were analyzed using IBM SPSS vn. 23 software. Conformity of the data to normal distribution was examined with skewness-kurtosis values. In the comparisons between the groups of the insulin application skill level points, which did not show normal distribution, the Kruskal Wallis test was used, and multiple comparisons were examined with the Dunn test. The Friedman test was applied to comparisons of the insulin application skill level points within groups and of different groups not showing normal distribution according to time. Multiple comparisons were examined with the Dunn test. Linear regression analysis was used in the examination of the effect of independent variables on the mid-test and final test points. Analysis results were stated as mean ± standard deviation (SD) or median (minimum-maximum) values for quantitative data, and as number (n) and percentage (%) for categorical data. A value of p<0.05 was accepted as the level of statistical significance and 95% as the confidence interval.

ELIGIBILITY:
Inclusion Criteria:

Nursing students Having completed all stages of the working process Not having received any insulin administration training before

Exclusion Criteria:

Not meeting the study inclusion criteria in full.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2024-02-15 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
Insulin skill 1nd measurement | One mounth
  insulin skill 1nd measurement

SECONDARY OUTCOMES:
Insulin skill 2nd measurement | Three mounth
  insulin skill 2nd measurement

CONTACTS AND LOCATIONS:
Locations (1):
- 1Kahramanmaraş Sütçü İmam University, Kahramanmaraş, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
The authors are unable or have chosen not to specify which data were used.

REFERENCES:
- [Derived] Soylu A, Seven A, Soylu D. The impact of training using six thinking hats versus video training on nursing students' insulin administration skills: a mixed-methods study. BMC Nurs. 2025 Jul 1;24(1):679. doi: 10.1186/s12912-025-03473-3. PMID 40598360
- See also: Related Info — https://doi.org/10.34087/cbusbed.1180986
- See also: Related Info — https://doi.org/10.24106/kefdergi.3150